CLINICAL TRIAL: NCT06677112
Title: Randomized Phase 3 Study of SELECTIVE SURGICAL STAGING Versus REFLEX Lymphadenectomy in Non-mappers Undergoing Sentinel Lymph Node Sampling for the Treatment of Endometrial Cancer
Brief Title: MCC-24-GYN-11: Comparison of Nodal Sampling in Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Miller (Other)
Responsible Party: Sponsor-Investigator, Rachel Miller, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98450
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer
Keywords: selective surgical staging; lymphadenectomy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Reflex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective Surgical Staging with side-specific lymphadenectomy (LAD) (Experimental): Pathologist and surgeon jointly perform the Intraoperative Consultation (IOC).
  Interventions: Procedure: Selective surgical staging
- REFLEX side-specific LAD (Active Comparator): Sentinel node procedure
  Interventions: Procedure: REFLEX

INTERVENTIONS:
Procedure: Selective surgical staging — Intraoperative Consultation, performed by pathologist and surgeon jointly. The uterus is inspected for extra-corpus spread (cervix, parametria, adnexa, distant). The surgical pathologist will evaluate the uterus according to the IOC Worksheet and promptly notify the surgeon of the results. The IOC will include evaluation for extra-corpus disease, lesion measurement, frozen section (to confirm measured lesion is malignant, cell type, and re-grading of tumor). Non-sentinel nodes will be handled according to institutional standard-of-care practice.
  Arms: Selective Surgical Staging with side-specific lymphadenectomy (LAD)
Procedure: REFLEX — The surgeon will perform a side-specific lymphadenectomy when there is no mapping on a hemipelvis (no tracer uptake in nodes). If neither side has successful Sentinel Node mapping, the surgeon performs a complete pelvic lymphadenectomy. Surgeons will remove the para-aortic lymph nodes at their discretion.
  Arms: REFLEX side-specific LAD

SUMMARY:
This study aims to estimate the recurrence-free survival rates in women with endometrial cancer treated with selective versus sentinel node surgical staging. This study will gather information to help determine the best way to evaluate lymph nodes during surgery for endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for complete hysterectomy and bilateral salpingooophorectomy with pelvic and aortic lymphadenectomy
* Histologically or cytologically confirmed carcinoma of the endometrium confined to the uterine corpus
* No clinical evidence of extra-uterine disease on pre-operative evaluation. Preoperative evaluation to rule-out extra-uterine disease may include a CT scan, MRI or ultrasound. Note: preoperative imaging is not mandatory for study enrollment.
* Prior systemic chemotherapy is allowed so long as it was at least five years prior to study enrollment, and there is no evidence of disease after such therapy.

Neoadjuvant chemotherapy for this endometrial cancer is not allowed.

* Life expectancy (estimated survival) of at least 6 months.
* AST(SGOT)/ALT(SGPT) < 3.0X upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* GOG Performance Status greater than 2 (Appendix II)
* Uterine sarcoma
* Clinical evidence of disease that extends beyond the uterus, including the presence of suspicious aortic or inguinal nodes on imaging or clinical exam
* Previous vaginal, pelvic or abdominal irradiation
* Chemotherapy or immunotherapy directed at the present disease
* Previous pelvic lymphadenectomy or retroperitoneal surgery
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen should be excluded
* Known allergy to iodine or indocyanine green (ICG) tracer, or allergic reactions to compounds of similar chemical or biologic composition
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women. Women of child-bearing potential will be excluded if they have a positive serum/urine pregnancy test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | up to 5 years
  Participants with no measurable disease from study entry until disease recurrence, death, or date of the last contact

SECONDARY OUTCOMES:
Concordance between selective surgical staging and final pathology Incidence | 5 years
  Percentage of participants for whom selective surgical staging and final pathology match
Progression-free survival | up to 5 years
  period from study entry until disease progression, death, or date of the last contact
Disease-specific Survival | up to 5 years
  period from study entry until death from the disease (endometrial cancer)
Overall patient survival rate | 5 years
  period from study entry until death from any cause

OTHER OUTCOMES:
Location patterns of nodal involvement associated with staging procedures | 5 years
Location patterns of nodal involvement associated with disease stage | 5 years
Patterns of nodal involvement associated with histological characteristics | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Miller, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No